CLINICAL TRIAL: NCT06020807
Title: Analytical Specificity of Bladder EpiCheck Test in Healthy Population and Urology Patients Without Prior History or Evidence of Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UC-Bladder EpiCheck-FDA-02
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Non Muscle Invasive Bladder Cancer; Non-Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy subjects and urology patients without prior history or evidence of bladder cancer
  Interventions: Diagnostic Test: Bladder EpiCheck

INTERVENTIONS:
Diagnostic Test: Bladder EpiCheck — Bladder EpiCheckTM (EpiCheck) is a urine test for monitoring of recurrence of NMIBC based on analysis of 15 informative DNA methylation biomarkers.

SUMMARY:
This is a prospective study to establish the analytical specificity of Bladder EpiCheck test in urine samples from healthy population and urology patients without prior history or evidence of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 or older
* Able to sign the informed consent form
* Normal, healthy subjects or subjects with one of the following conditions:

  1. Benign non-genitourinary disease (e.g. heart disease)
  2. Non-genitourinary cancers (e.g. lung, CRC, breast)
  3. Genitourinary disease other than bladder cancer including:
  4. Benign prostatic hyperplasia (BPH)
  5. Microhematuria proven negative for bladder cancer through prior UCC evaluation
  6. Inflammation/infection
  7. Symptomatic sexually transmitted disease (STD)
  8. Urinary tract stones
  9. Genitourinary trauma
* Subjects with native bladder

Exclusion Criteria:

* Known current or prior diagnosis of bladder cancer (non-muscle or muscle invasive)
* Currently in work-up due to suspicion of cancer of any kind

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and urology patients without prior history or evidence of bladder cancer will be recruited from urology group clinics.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Specificity | Day 1
  The primary endpoint of the study is the specificity of the Bladder EpiCheck Test in healthy population.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No